CLINICAL TRIAL: NCT01149304
Title: Evaluation of the Preventive Effect of Enoxaparin, Pentoxifylline and Ursodeoxycholic Acid to Radiation Induced Liver Toxicity After Brachytherapy of Liver Metastases From Colorectal Carcinoma, Assessed in a Prospective Randomised Trial
Brief Title: Preventive Effect of Enoxaparin, Pentoxifylline and Ursodeoxycholic Acid to Radiation Induced Liver Toxicity
Acronym: ELDORADO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Principal Investigator, Robert Damm, Dr. med. Robert Damm, University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAD052; 2008-002985-70 (EudraCT Number); MD-R20080507 (Other: Sponsor's protocol code number)
Record Dates: First submitted 2010-06-04; First posted 2010-06-23 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Cancer; Liver Metastases; Irradiation Damage; Radiation Induced Liver Disease
Keywords: brachytherapy; liver metastases; irradiation; radiation induced liver disease; dosimetry
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pentoxifylline; Ursodeoxycholic Acid; Enoxaparin

ARMS (2):
- Group A (Experimental): Medication group with patients receiving the study medication according to the study protocol for 8 weeks after HDR brachytherapy.
  Interventions: Drug: Pentoxifylline; Drug: Ursodeoxycholic Acid; Drug: Enoxaparin
- Group B (No Intervention): Comparison group with patients receiving the standard therapy of HDR brachytherapy without the study specific medication.

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline is given for 8 weeks since the evening of the day of intervention with a dose of 400mg applied three times daily (morning, noon, evening).
  Other Names: Trental (CAS 6493-05-6, ATC C04AD03)
  Arms: Group A
Drug: Ursodeoxycholic Acid — Ursodeoxycholic acid is administered for 8 weeks since the evening of the day of intervention. Dosage is 250mg given three times daily (morning, noon, evening).
  Other Names: Ursofalk (CAS 128-13-2, ATC A05AA02)
  Arms: Group A
Drug: Enoxaparin — Enoxaparin with a dose of 40mg is injected subcutaneously once a day for 8 weeks since the evening of the day of intervention after the HDR-brachytherapy.
  Other Names: Clexane (CAS 9005-49-6, ATC B01AB05)
  Arms: Group A

SUMMARY:
To evaluate whether a combination regimen of pentoxifylline, ursodeoxycholic acid and enoxaparin provides a protective effect on the liver parenchyma after high dose rate (HDR) brachytherapy.

DETAILED DESCRIPTION:
A preventive effect of pentoxifylline, ursodeoxycholic acid and low dose low molecular weight heparin on pathological processes in healthy tissue after irradiation is described in clinical studies on percutaneous liver irradiation and on bone marrow transplantation. However, data remains inconclusive.

This exploratory study aims at assessing whether a protective effect of the combination of pentoxifylline, ursodeoxycholic acid and enoxaparin can be demonstrated in a limited number of patients with liver metastases of colorectal cancer after HDR brachytherapy.

All patients receive a single fraction CT/MRI-guided HDR-brachytherapy of colorectal liver metastases using Iridium-192 as a standard therapy. The follow-up consists of 4 MRI controls of the abdomen using the hepatocyte-specific contrast agent Gd-EOB-DTPA (Primovist) after 3 days, 6 weeks, 3 months and 6 months as well as blood samples and a questionnaire taken the same time.Within the study, 22 patients are given low dose low molecular weight heparin, pentoxifylline and ursodeoxycholic acid for 8 weeks starting with the preinterventional day. Another 22 patient will receive the standard therapy without the medication. After completion of the follow-up, MRI volume data of the lesion will be acquired and compared to the dosimetric treatment plan. Blood samples are tested for liver-specific and inflammatory laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* If female, postmenopausal or surgically sterilized
* Liver metastases from colorectal carcinoma scheduled for a CT/MRI-guided single-fraction interstitial HDR brachytherapy
* Non-cirrhotic liver
* Life expectancy longer than 6 months
* willing and able to undergo all study procedures
* Having voluntarily provided written and fully informed consent

Exclusion Criteria:

* Women who are pregnant, lactating or who are of childbearing potential
* Liver cirrhosis
* Hepatitis B
* Hepatitis C
* Patients being clinically unstable
* Uncooperative, in the investigator's opinion
* Having been previously enrolled in this study
* Participating in another therapy-modulating clinical trial
* Contraindication for MRI
* Contraindication or hypersensitivity to one or more components of Gd-EOB-DTPA, Enoxaparin, Ursodeoxycholic acid and/or Pentoxifylline
* Any prior irradiation therapy of the liver
* Close affiliation with the investigational site; e.g. a close relative of the investigator
* Severe coronary artery disease
* Autoimmune diseases
* Acute bacterial endocarditis
* Active major bleedings and high rish of uncontrolled haemorrhage
* Patients with severe or moderate renal impairment (GFR below 60 mL/min/1.73 m2 according to the MDRD or Cockroft-Gault formula, calculated from a creatinine value obtained within 1 week before each planned Primovist-enhanced MR examination)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
HDR-brachytherapy isodose (measured in Gy) that corresponds to the metastases without enhancement of Gd-EOB-DTPA in MR imaging using an axial T1 THRIVE sequence. | One day prior to brachytherapy.
  The primary variable is the HDR-brachytherapy isodose that encloses liver tissue with a diminished uptake of the hepatocyte selective contrast agent GD-EOB-DTPA. By identifying the damaged volume in every layer of the axial T1 THRIVE image, 3D data can be calculated and correlated to a specific isodose when merged with the 3D irradiation treatment plan.
  Prior to brachytherapy, the baseline volume of the metastases will be measured instead of the liver tissue damaged by irradiation.
HDR-brachytherapy isodose (measured in Gy) that corresponds to the irradiated liver tissue without enhancement of Gd-EOB-DTPA in MR imaging using an axial T1 THRIVE sequence. | 3 days after brachytherapy.
  The primary variable is the HDR-brachytherapy isodose that encloses liver tissue with a diminished uptake of the hepatocyte selective contrast agent GD-EOB-DTPA. Liver tissue without enhancement of Gd-EOB-DTPA around the irradiated metastases is defined as damaged by irradiation.
  By identifying the irreversibly damaged volume in every layer of the axial T1 THRIVE image, 3D data can be calculated and correlated to a specific isodose when merged with the 3D irradiation treatment plan.
  Imaging up to 3 months after brachytherapy is mandatory for inclusion in the analysis.
HDR-brachytherapy isodose (measured in Gy) that corresponds to the irradiated liver tissue without enhancement of Gd-EOB-DTPA in MR imaging using an axial T1 THRIVE sequence. | 6 weeks after brachytherapy.
  The primary variable is the HDR-brachytherapy isodose that encloses liver tissue with a diminished uptake of the hepatocyte selective contrast agent GD-EOB-DTPA. Liver tissue without enhancement of Gd-EOB-DTPA around the irradiated metastases is defined as damage by irradiation.
  By identifying the irreversibly damaged volume in every layer of the axial T1 THRIVE image, 3D data can be calculated and correlated to a specific isodose when merged with the 3D irradiation treatment plan.
  Imaging up to 3 months after brachytherapy is mandatory for inclusion in the analysis.
HDR-brachytherapy isodose (measured in Gy) that corresponds to the irradiated liver tissue without enhancement of Gd-EOB-DTPA in MR imaging using an axial T1 THRIVE sequence. | 3 months after brachytherapy.
  The primary variable is the HDR-brachytherapy isodose that encloses liver tissue with a diminished uptake of the hepatocyte selective contrast agent GD-EOB-DTPA. Liver tissue without enhancement of Gd-EOB-DTPA around the irradiated metastases is defined as damage by irradiation.
  By identifying the irreversibly damaged volume in every layer of the axial T1 THRIVE image, 3D data can be calculated and correlated to a specific isodose when merged with the 3D irradiation treatment plan.
  Imaging up to 3 months after brachytherapy is mandatory for inclusion in the analysis.
HDR-brachytherapy isodose (measured in Gy) that corresponds to the irradiated liver tissue without enhancement of Gd-EOB-DTPA in MR imaging using an axial T1 THRIVE sequence. | 6 months after brachytherapy.
  The primary variable is the HDR-brachytherapy isodose that encloses liver tissue with a diminished uptake of the hepatocyte selective contrast agent GD-EOB-DTPA. Liver tissue without enhancement of Gd-EOB-DTPA around the irradiated metastases is defined as damage by irradiation.
  By identifying the irreversibly damaged volume in every layer of the axial T1 THRIVE image, 3D data can be calculated and correlated to a specific isodose when merged with the 3D irradiation treatment plan.
  Imaging up to 3 months after brachytherapy is mandatory for inclusion in the analysis.

SECONDARY OUTCOMES:
Correlation between the HDR brachytherapy isodose that corresponds to damaged live tissue as defined by missing Gd-EOB-DTPA enhancement in MR imaging and liver-specific laboratory values. | One day prior to brachytherapy, 3 days, 6 weeks, 3 months and 6 months after brachytherapy.
  To evaluate the relation between hepatocyte dysfunction by irradiation as assessed in GD-EOB-DTPA-enhanced MRI and changes in liver-specific and inflammatory laboratory values.
  The following laboratory values are included:
  * bilirubin
  * ASAT/ALAT
  * albumin
  * ChE
  * gamma-GT
  * GLDH
  * INR
  * fibrinogen
  * fibrin monomer
  * factor VIII
  * IL 2 + 6
  * PAI
  * protein c + s
  * vWF
  * AT3
Quality of live. | One day prior to brachytherapy, 3 days, 6 weeks, 3 months and 6 months after brachytherapy.
  To evaluate the quality of live comparing both patient groups using the EQ-5D questionnaire and ECOG performance status.
Safety of the study drugs. | Up to 6 months after brachytherapy.
  To assess the safety of the combination regimen of pentoxifylline, low dose low molecular weight heparin, and ursodeoxycholic acid given after HDR brachytherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ricke, MD — University of Magdeburg, Faculty for Medicine; Robert Damm, MD, Principal Investigator — University of Magdeburg, Faculty for Medicine
Locations (1):
- Clinic for Radiology and Nuclear Medicine, Magdeburg, Saxony-Anhalt, Germany

REFERENCES:
- [Result] Seidensticker M, Seidensticker R, Damm R, Mohnike K, Pech M, Sangro B, Hass P, Wust P, Kropf S, Gademann G, Ricke J. Prospective randomized trial of enoxaparin, pentoxifylline and ursodeoxycholic acid for prevention of radiation-induced liver toxicity. PLoS One. 2014 Nov 13;9(11):e112731. doi: 10.1371/journal.pone.0112731. eCollection 2014. PMID 25393877